CLINICAL TRIAL: NCT06327802
Title: Improving the Well-being of Caregivers of Cystic Fibrosis Patients During Physiotherapy Treatment
Acronym: MucoZar
Status: Recruiting | Type: Observational
Sponsor: Pole Sante Grace de Dieu (Other)
Responsible Party: Sponsor
Other Study IDs: 20240104
Record Dates: First submitted 2024-03-17; First posted 2024-03-25 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; caregivers; burden
MeSH Terms: conditions — Cystic Fibrosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Participants will have to answer the socio-demographic questions (Age, weight, height, FEV1, FVC) and the Beck, Zarit, HAD, FAS CARERQOL-7D questionnaires

SUMMARY:
The main objective of the study is to determine the impact of cystic fibrosis affecting a child on the parents' quality of life, their possible anxiety and depressive symptoms, their general fatigue and the feeling of burden in these caregivers.

DETAILED DESCRIPTION:
Cystic fibrosis is the most common rare genetic disease in France, and in European countries in general. According to current epidemiological data, 80,000 people worldwide are affected. It represents a major public health issue, as it is a chronic disease that has a major impact on the life expectancy of affected patients. Thanks to the latest medical advances, promising treatments are now available, helping to improve patient survival rates to over 40-50 years. Among existing treatments, respiratory and musculoskeletal physiotherapy are highly recommended. It will play a key role throughout the life of a cystic fibrosis patient. Patients with chronic respiratory diseases are at high risk of developing anxiety and depressive symptoms. As the disease worsens, the patient becomes increasingly dependent, leading to restrictions in participation and activities of daily living. As a result, the presence of family and friends is of paramount importance in ensuring that sick children adhere to treatment and take their medication. However, this workload on the part of a parent, who has to make major changes to their lifestyle in order to adapt to their child's treatment, can have a considerable impact on their well-being, and increase the risk of anxiety/depression, even leading to burnout. Psychologists have studied the subject of assessing quality of life in parents of children with cystic fibrosis. At present, knowing that the quality of life of sufferers is as much affected as that of their caregivers, questionnaires have been introduced to assess parents' quality of life, notably the CarerQol-7D . The aim of this study would be to raise the issue of exhaustion among parents of children with cystic fibrosis, and to consider how to reduce the impact of this heavy mental burden on them. This would contribute to better therapeutic adherence and improved treatment of children. To this end, questionnaires and interviews could be set up with parents, with the aim of developing a relevant and optimal action strategy for their children.

ELIGIBILITY:
Inclusion Criteria:

* parents (father, mother, dyads (father+mother) of children suffering from cystic fibrosis) who agree to answer the various questionnaires.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects recruited are parents (father, mother, dyads (father+mother) of children suffering from cystic fibrosis) who agree to answer the various questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Zarit Burden Interview | 1 year
  The Zarit Burden Interview, a popular caregiver self-report measure used, contains 22 items. Each item on the interview is a statement which the caregiver is asked to endorse using a 5-point scale. Response options range from 0 (Never) to 4 (Nearly Always).

CONTACTS AND LOCATIONS:
Locations (1):
- PSLA GDD, Caen, France

IPD SHARING:
Plan to Share IPD: No